CLINICAL TRIAL: NCT05268913
Title: Robust EArly Detection of bReast Cancer in hIgh riSK Premenopausal Population Using Novel Lipid Based Imaging Methods
Brief Title: Towards Early Detection of Breast Cancer in High Risk Population
Acronym: READ RISK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-102-21
Record Dates: First submitted 2022-02-14; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with BRCA1/2 genes
  Interventions: Diagnostic Test: MRI scan; Biological: Blood test
- Women with breast cancer
  Interventions: Diagnostic Test: MRI scan; Biological: Blood test
- Women with obesity
  Interventions: Diagnostic Test: MRI scan; Biological: Blood test

INTERVENTIONS:
Diagnostic Test: MRI scan — Participants will undertake a magnetic resonance imaging scan.
Biological: Blood test — Participants will undertake a fasting blood test.

SUMMARY:
Breast cancer is a major and growing health challenge, and the leading cause of cancer in women. As population obesity rates increase, the number of new breast cancer diagnosis continues to rise. Despite treatment advances, breast cancer remains an important cause of premature mortality, taking women in the prime of life. Although underlying susceptibility caused by mutation in the genes including BRCA1/2 is increasingly identified, current pre-symptomatic screening for the general population and those at high genetic risk remains sub-optimal, with high false negative and positive rates.

Alteration of breast lipid composition has been observed by us and others in patients with breast cancer and is thought to precede onset. We have developed and tested a novel method to allow a standard 3T MRI scanner to perform quantitative 3D mapping of specific lipid molecules in the breast.

We will investigate if this method can detect very early breast cancers, and compare the amount and spread of lipid composition in breast tissue of premenopausal women with very high genetic risk of breast cancer, women with breast cancer and women with obesity.

ELIGIBILITY:
Inclusion Criteria:

-

Women with BRCA1/2 genes:

* female 18-55 years old, premenopausal
* BRCA 1/2 gene carriers
* not having any metabolic disorders (e.g., diabetes)
* not on any long term medications that may affect lipid metabolism (e.g., statins)
* BMI < 30

Women with breast cancer (no obesity):

* females 18-55 years old, premenopausal
* confirmed diagnosis of invasive ductal carcinoma of the breast
* not having any metabolic disorders (e.g., diabetes)
* not on any long term medications that may affect lipid metabolism (e.g., statins)
* BMI < 30

Women with breast cancer (obesity):

* BMI > 30
* otherwise as women with breast cancer

Women with obesity:

* females 18-55 years old, premenopausal
* not having any metabolic disorders (e.g., diabetes)
* not on any long term medications that may affect lipid metabolism (e.g., statins)
* BMI > 30

Exclusion Criteria:

* females under 18 or over 55 years old, postmenopausal
* males
* have metabolic disorders (e.g., diabetes)
* on long term medications that may affect lipid metabolism (e.g., statins)
* contraindicated for MR investigation (poor renal function and metal implants)
* (for patients) concurrent cancer in other sites
* (for patients) started hormone treatment, chemotherapy or breast surgery
* non-English speakers

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with BRCA1/2 genes will be identified and approached by the geneticist and research nurse at the family high risk clinic. Patients will be identified and approached by the breast surgeon and breast care nurse at the results clinic. Women with obesity will be identified through organisation emails, word of month and leaflets in the community health clinic for residents of Aberdeenshire.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Amount of lipid composition in the breast | One hour
  The percentage of monounsaturated fatty acids, polyunsaturated fatty acids and saturated fatty acids relative to total lipid will be measured using magnetic resonance imaging (MRI) scanner software and MATLAB computer programme.
  Unit of Measurement: %.
Spatial distribution (skewness) of lipid composition in the breast | One hour
  Skewness measures the asymmetry in distribution. The skewness of lipid composition in the breast will be measured using MRI scanner software and MATLAB computer programme.
  Unit of Measurement: unitless.
Spatial distribution (entropy) of lipid composition in the breast | One hour
  Entropy measures the randomness in distribution. The entropy of lipid composition in the breast will be measured using MRI scanner software and MATLAB computer programme.
  Unit of Measurement: unitless.
Spatial distribution (kurtosis) of lipid composition in the breast | One hour
  Kurtosis measures the peakedness in distribution. The kurtosis of lipid composition in the breast will be measured using MRI scanner software and MATLAB computer programme.
  Unit of Measurement: unitless.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Biomedical Imaging Centre, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No